CLINICAL TRIAL: NCT04463511
Title: Placing Preterm Infants in Polyethylene Bags Immediately After Birth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Dublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: APOLLO_PB_BCC
Record Dates: First submitted 2020-07-03; First posted 2020-07-09 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Newborn; Infant; Hypothermia; Premature
Keywords: cord clamping; hypothermia; hyperthermia; polyethylene bag
MeSH Terms: conditions — Hypothermia; Premature Birth; Hyperthermia

STUDY DESIGN:
Intervention Model Description: Single-centre randomised controlled trail
Who Masked: Participant, Outcomes Assessor
Masking Description: In the delivery room, the infant is randomised to application of a polyethylene bag before or after cord clamping. Neither the delivery room care provider nor the investigator are blinded to the group assignment. When the infant is stable, they are be transferred from the delivery room to the neonatal unit. The outcome assessor is the admitting nurse in the neonatal unit who will be blinded to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PB BCC: Polyethylene Bag Before Cord Clamping (Experimental): Immediately after delivery, while still attached to placental circulation, infants will be placed in a PB. After the cord has been clamped and cut, the infant will be transferred to the resuscitaire for ongoing care. In the case of caesarean section a sterile bag will be used and prepared observing sterile techniques. A member of the neonatal team donned in sterile gown and gloves will assist the obstetrician in placing the infant in the PB.
  Interventions: Other: Polyethylene bag before the umbilical cord is clamped
- PB ACC: Polyethylene Bag After Cord Clamping (No Intervention): Infants will not be placed in a PB immediately after birth. After the cord has been clamped and cut, the infant will be transferred to the resuscitaire where they will be placed in a PB.

INTERVENTIONS:
Other: Polyethylene bag before the umbilical cord is clamped — 11" x 16" (279mm x 406mm) sterile resealable PB (Resealable Polybag, Helapet Ltd, Bedfordshire, UK)
  Arms: PB BCC: Polyethylene Bag Before Cord Clamping

SUMMARY:
Primary objective: To determine if placing preterm infants in a polyethylene bag (PB) immediately after birth, before the umbilical cord is clamped, will increase the number of preterm infants with a normal temperature on admission to the Neonatal Intensive Care Unit (NICU).

DETAILED DESCRIPTION:
Newly born preterm infants that develop abnormal temperature after birth have higher morbidity and mortality. Placing infants < 32 weeks' gestation in a polyethylene bag (PB) in the delivery room (DR) reduces the rate of hypothermia on admission to the Neonatal Intensive Care Unit (NICU). Since 2012, the rate of admission hypothermia in preterm infants, placed in a PB in the DR at the National Maternity Hospital (NMH), has increased significantly. This may be as a result of heat loss while the infant remains attached to the cord.

Our primary objective is to determine if placing preterm infants in a PB immediately after birth, before the umbilical cord is clamped will increase the number of preterm infants with a normal temperature on admission to the NICU.

ELIGIBILITY:
Inclusion Criteria:

Infants who are inborn at the National Maternity Hospital at < 32 (up to 31+6) weeks' gestation by best obstetric estimate will be included in the study.

Exclusion Criteria:

* Infants with a large abdominal wall or neural tube defects
* Infants with an imperforate anus
* Infants to whom resuscitative measures are not initiated in the DR

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 194 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Temperature on admission to the Neonatal Intensive Care Unit (NICU) | The primary outcome measure will be determined on admission to the NICU, before the infant is removed from the transport incubator (< 90minutes of life)
  Rectal temperature recorded upon arrival to the NICU, while the infant is in the transport incubator. (measured in degrees celsius)

SECONDARY OUTCOMES:
Respiratory support in the DR | Within 2 hours of birth
  Type and duration of respiratory support in the DR
5 minute Apgar | Within 2 hours of birth
  Scale (0-10)
External cardiac massage in the delivery room | Within 2 hours of birth
  Yes/ No, Duration
Infant temperature recordings in the delivery room | Within 2 hours of birth
  Measured with Microlife MT 1931 digital thermometer at the rectum. Recorded in degrees celsius.
Axillary temperature on admission to the NICU | Between 0-2 hours of life
  Measured with Microlife MT 1931 digital thermometer at the rectum. Recorded in degrees celsius.
Temperature 1 hour after admission | Between 0-2 hours of life
  Measured with Microlife MT 1931 digital thermometer at the rectum. Recorded in degrees celsius.
Central catheter placement in first 24 hours | Between 0-24 hours of life
  Yes/no. Type and location of catheter
Intubation and mechanical ventilation | Term corrected gestation age or hospital discharge (<17 weeks)
  Yes/no, type and duration
Respiratory Distress Syndrome | Between 0-24 hours of life
  Yes/no
Non-invasive ventilation (NIV) on the first day of life (24 hours) | Between 0-24 hours of life
  Yes/ no, type of NIV
Surfactant administration | Day 1 - 7 of life
  Yes/ no, route of administration
Pneumothorax requiring drainage | Term corrected gestation age or hospital discharge (<17 weeks)
  Yes/ no, needle aspiration or definitive chest drain or both
Pulmonary haemorrhage | Term corrected gestation age or hospital discharge (<17 weeks)
  Yes/ no
Hypotension requiring inotropes | Term corrected gestation age or hospital discharge (<17 weeks)
  Yes/ no, inotropes, duration
Intraventricular haemorrhage | Term corrected gestation age or hospital discharge (<17 weeks)
  Papile classification
Periventricular leukomalacia | Term corrected gestation age or hospital discharge (<17 weeks)
  Yes/ no
Necrotising enterocolitis | Term corrected gestation age or hospital discharge (<17 weeks)
  Bell's staging criteria
Sepsis - early onset | Between 0-72 hours of life
  Yes/ no
Sepsis - late onset | After 72 hours of life until term corrected or hospital discharge (maximum 16 weeks)
  Yes/ no
Retinopathy of prematurity requiring treatment | Term corrected gestation age or hospital discharge (<17 weeks)
  Yes/ no, treatment
Oxygen requirement at 36 weeks corrected gestational age | 36 weeks corrected gestational age
  Yes/ no
Death before discharge from hospital | Term corrected gestation age or hospital discharge (<17 weeks)
  Yes/ no

CONTACTS AND LOCATIONS:
Overall Officials: Lisa K McCarthy, MB BCh BAO, Principal Investigator — National Maternity Hospital / University College Dublin
Locations (1):
- National Maternity Hospital, Dublin, Dubiln, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McCall EM, Alderdice F, Halliday HL, Vohra S, Johnston L. Interventions to prevent hypothermia at birth in preterm and/or low birth weight infants. Cochrane Database Syst Rev. 2018 Feb 12;2(2):CD004210. doi: 10.1002/14651858.CD004210.pub5. PMID 29431872
- [Result] Laptook AR, Salhab W, Bhaskar B; Neonatal Research Network. Admission temperature of low birth weight infants: predictors and associated morbidities. Pediatrics. 2007 Mar;119(3):e643-9. doi: 10.1542/peds.2006-0943. Epub 2007 Feb 12. PMID 17296783
- [Derived] Dunne EA, Ni Chathasaigh CM, Geraghty LE, O'Donnell CP, McCarthy LK. Polyethylene bags before cord clamping in very preterm infants: a randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2024 Apr 18;109(3):317-321. doi: 10.1136/archdischild-2023-325808. PMID 38212105